CLINICAL TRIAL: NCT07060599
Title: A Prospective Multicenter Randomized Trial Comparing the Human-AI Collaborative INSIGHT Workflow vs. Conventional Pathology Diagnosis for Detecting Invasive Carcinoma in Breast Cancer With Extensive Intraductal Component (EIC)
Brief Title: Human-AI Collaborative INSIGHT Diagnostic Workflow for in Breast Cancer With Extensive Intraductal Component
Acronym: INSIGHT-EIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Peng Sun, MD, PhD, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: G2023-277-01
Record Dates: First submitted 2025-06-24; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Artificial Intelligence (AI) in Diagnosis
Keywords: Extensive Intraductal Component; Breast Cancer; Pathology; Human-AI Collaborative Workflow; Artificial Intelligence; DCIS; Diagnosis
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Workflow (No Intervention): Pathologists review all WSIs without AI assistance; IHC stains ordered at pathologist's discretion.
- INSIGHT Workflow (Experimental): AI pre-screening of WSIs; AI-generated ROI maps highlighting suspicious invasive cancer regions; Pathologist verifies AI-flagged ROIs and full slide review; IHC only triggered for uncertain ROIs if necessary.
  Interventions: Other: INvasion Screening with Intelligent Guidance for Histopathology Triage (INSIGHT) Workflow

INTERVENTIONS:
Other: INvasion Screening with Intelligent Guidance for Histopathology Triage (INSIGHT) Workflow — An AI-generated segmentation model are refined through a post-processing pipeline: retaining only invasive carcinoma (IC) regions, filtering detections <500 µm², grouping adjacent IC areas, and generating per-cluster bounding boxes (red boxes). This converted raw segmentations into clinically actionable ROI proposals, balancing sensitivity and specificity for pathologist review in external testing and clinical validation. The INSIGHT workflow addresses key diagnostic challenges in EIC cases by pre-screening whole-slide images (WSIs) and intelligently marking potential IC regions. This guides pathologists to prioritize diagnostically critical areas across multiple slides or within extensive DCIS - a task particularly valuable when IC is multifocal or presents as subtle micro-invasive foci easily overlooked during routine manual examination.
  Arms: INSIGHT Workflow

SUMMARY:
The goal of this clinical trial is to see if an artificial intelligence (AI)-assisted method helps doctors more accurately detect invasive breast cancer in people with a specific type of tumor called "extensive intraductal carcinoma" (EIC). This type of tumor is challenging to diagnose correctly using standard methods. The main question this study aims to answer is: Does the new AI-assisted method find more invasive breast cancer in EIC tumors compared to the standard method?

Researchers will compare two groups:

* Group 1 (INSIGHT): Doctors review breast tissue samples using an AI tool that highlights suspicious areas needing closer attention.
* Group 2 (Conventional): Doctors review breast tissue samples without AI help, using the standard method.

This comparison will show if the AI-assisted method works better at finding invasive cancer.

What happens in the study?

* Researchers will use stored breast tissue samples already collected during the participant's surgery.
* Each sample will be randomly assigned to be reviewed using either the new AI-assisted method (Group 1) or the standard method (Group 2).
* In Group 1, an AI program will scan the tissue images first and point out areas that might contain invasive cancer for the doctor to check closely.
* In Group 2, doctors will review the tissue images without any AI help, using their standard process.
* Researchers will measure which method finds invasive cancer more accurately, how long the review takes, and how many additional tests (called IHC stains) are needed.

No new procedures are required from participants; the study uses existing tissue samples.

DETAILED DESCRIPTION:
Breast cancer with extensive intraductal component (EIC) presents significant diagnostic challenges, characterized by widespread ductal carcinoma in situ (DCIS) frequently accompanied by small invasive foci (≤10 mm). Accurate identification of invasive carcinoma in EIC is critical for clinical staging and treatment decisions, yet conventional diagnostic methods face substantial limitations. Pathologists must manually screen extensive DCIS regions for minute invasive components, a labor-intensive process with reported miss rates reaching 20%, particularly for microinvasive foci (≤1 mm). Diagnostic uncertainty frequently leads to excessive immunohistochemical (IHC) staining (e.g., p63, CK5/6), with each stain costing ¥373.40, significantly increasing healthcare costs and prolonging turnaround times.

To address these challenges, we developed the INSIGHT (INvasion Screening with Intelligent Guidance for Histopathology Triage) human-AI collaborative workflow. This solution integrates four public datasets (TiGER, BRACS, BACH, CAS_PUIH) and employs weakly supervised pseudo-labeling to expand annotated pixels 22-fold to 25 billion, specifically improving representation of DCIS (3.14% to 12.53%) and benign tissue (0.65% to 10.9%). The AI model, based on a UperNet-VAN architecture, achieved Dice scores of 0.877 (training), 0.853 (validation), and 0.847 (testing). The system processes segmented invasive regions through size filtering (>500 µm²) and cluster grouping to generate actionable regions of interest (ROIs) for pathologist guidance.

In our preliminary retrospective study (576 whole slide images from 44 EIC patients), the INSIGHT workflow demonstrated superior diagnostic performance compared to conventional methods: sensitivity improved from 82.7% to 95.1% (p<0.001), with particularly notable gains in detecting ≤1 mm microinvasive foci (69.4% to 91.8%); negative predictive value (NPV) reached 96.7% versus 89.6% (p<0.001). The workflow reduced mean diagnostic time by 41.4% (102.6 to 60.1 seconds per slide, p<0.001) and decreased IHC usage by 40.4% (p=0.011). While standalone AI showed high sensitivity (95.6%), its specificity remained limited (76.6%), underscoring the necessity of human-AI collaboration.

This prospective clinical trial aims to validate the INSIGHT workflow's generalizability in real-world clinical settings, quantify its impact on patient stratification and treatment decisions, and establish standardized protocols for AI-assisted diagnosis to bridge critical gaps in computational pathology translation from research to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* DCIS (ductal carcinoma in situ) with or without invasive carcinoma, as confirmed by core needle biopsy prior to surgery.
* Tumor size >2 cm (cT2-cT4 according to AJCC 8th edition staging) with extensive calcifications, as documented by ultrasound or MRI.
* Undergone either mastectomy or breast-conserving surgery.
* Histopathological examination showing DCIS comprising ≥80% of the total tumor volume in the surgical specimen.

DCIS (ductal carcinoma in situ) with or without invasive carcinoma, as confirmed by core needle biopsy prior to surgery.

- Minimum of 10 H&E-stained slides available for each case, with adequate tissue quality for analysis.

Exclusion Criteria:

* Received neoadjuvant therapy (chemotherapy, endocrine therapy, or targeted therapy) before surgery.
* History of vacuum-assisted biopsy (VAB) or other minimally invasive breast procedures that may alter tumor architecture.
* Insufficient or degraded tissue samples (e.g., due to fixation artifacts, sectioning errors, or poor staining quality).
* Tumors lacking a DCIS (ductal carcinoma in situ) component upon histological examination.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 480 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic sensitivity | through study completion, an average of 1 year
  Diagnostic sensitivity for invasive carcinoma detection in breast cancer with extensive intraductal component

SECONDARY OUTCOMES:
Diagnostic efficiency | up to 24 weeks
  Diagnostic time cost per case (minutes)
Immunohistochemical (IHC) stains utilization | up to 24 weeks
  Immunohistochemical (IHC) stains utilization rate (stains/case)
Diagnostic specificity | through study completion, an average of 1 year
  Diagnostic specificity for invasive carcinoma detection in breast cancer with extensive intraductal component
Negative predictive value (NPV) | through study completion, an average of 1 year
  Negative predictive value (NPV) for invasive carcinoma detection in breast cancer with extensive intraductal component

CONTACTS AND LOCATIONS:
Overall Officials: Peng Sun, MD, PhD., Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No